CLINICAL TRIAL: NCT03036475
Title: Sentinel Lymph Node Biopsy Using a Magnetic Tracer Versus Standard Radio-isotope Technique in Early Breast Cancer
Brief Title: Sienna and Sentimag in Sentinel Lymph Node Biopsy
Acronym: Sienna
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yolanda Chan (Other)
Responsible Party: Sponsor-Investigator, Yolanda Chan, Associate Consultant, Kwong Wah Hospital
Organization: Kwong Wah Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 107-15
Record Dates: First submitted 2017-01-26; First posted 2017-01-30 (Estimated); Last update posted 2017-02-16 (Actual); Status verified 2017-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: Sienna+ injection — Subcutaneous injection of Sienna+ in the morning of operation day

SUMMARY:
The aim of this study is to evaluate a new method for the localization of breast cancer sentinel lymph node using Sienna+® and Sentimag® detection in comparison to our standard techniques with radio-isotopes.

DETAILED DESCRIPTION:
The use of radioisotope with or without blue dye has long become the gold standard for sentinel lymph node localization in the management of breast cancer. The latest evidence from a number of European trials has proven that a new tracer agent, superparamagnetic iron oxide particles (SPIOs, Sienna+®), is non-inferior to the standard method of lymphatic mapping. Its application and feasibility has yet been tried in most Asian countries.

This is a prospective paired comparison trial involving both the new magnetic technique and the standard method. Patients with preoperative diagnosis of invasive carcinoma or ductal carcinoma in-situ of the breast undergoing SNOLL (Sentinel node and occult lesion localization) will be recruited from the Breast Centre of Kwong Wah Hospital. Informed consent will be obtained. All patients recruited will receive subcutaneous injection of 2 ml of Sienna+® diluted with saline to 5 ml at Breast Centre in the morning of operation, followed by five minutes of massage to the injection site. Before incision, on-table transcutaneous detection with the handheld magnetometer are carried out after at least 20 minutes from injection. Intraoperative counts of sentinel lymph nodes identified as well as the ex-vivo counts of excised nodes are also measured. All procedures are supplemented with localization by radioisotope. All lymph nodes excised will be sent for histopathological examination.

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with early-stage breast cancer (including ductal carcinoma in-situ) who are clinically or radiologically node-negative and consenting for sentinel lymph node biopsy
* Patients undergoing SNOLL (Sentinel node and occult lesion localization) with the use of radio-isotope in our Breast Centre

Exclusion Criteria:

* Patients with clinically T3 or T4 breast cancer and any contraindication to sentinel lymph node biopsy
* Patients with pacemaker or other implantable device in the chest wall

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2017-03-01 (Estimated); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of successful procedures for sentinel lymph node identification (identification rate per patient) by the magnetic method compared with the standard method | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Yolanda Chan, MBBS, Principal Investigator — Kwong Wah Hospital

IPD SHARING:
Plan to Share IPD: No